CLINICAL TRIAL: NCT03980457
Title: Effects of Exoskeleton-Assisted Gait Training on Functional Rehabilitation Outcomes in Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10742
Record Dates: First submitted 2019-05-02; First posted 2019-06-10 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Weakness of Extremities as Sequela of Stroke
Keywords: Stroke; leg weakness; Exoskeleton
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Open label pragmatic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Exo-group (Experimental): Standard rehabilitation plus use of Exoskeleton
  Interventions: Device: Indego Exoskeleton; Other: Standard Rehabilitation
- Control-Group (Placebo Comparator): Standard rehabilitation
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Device: Indego Exoskeleton — Powered generated orthosis
  Arms: Exo-group
Other: Standard Rehabilitation — Standard Rehabilitation

SUMMARY:
The goal of this study is to determine the efficacy of electromechanical exoskeleton-assisted gait training on rehabilitation functional outcomes in patients with stroke undergoing therapy in an in-patient rehabilitation facility.

DETAILED DESCRIPTION:
Abstract

Objective: The goal of this study is to determine the efficacy of electromechanical exoskeleton-assisted gait training on rehabilitation functional outcomes in patients with stroke undergoing therapy in an in-patient rehabilitation facility.

Background:

Method: The investigators will study 50 patients with stroke consecutively admitted to a designated stroke rehabilitation unit in the Oklahoma City VA Medical Center. All patients will receive their daily 3-hours conventional therapy, plus an hour of either exoskeleton or over-ground gait training 3 times per week for 60 minutes. Patients were assigned to either the experimental (exoskeleton) or the control (over-ground) groups by computer-generated randomization. This is an open-label pragmatic trial, where neither the patients nor the clinicians could be masked to the intervention. Institution review board (IRB) approval will be obtained for the protocol. The demographic data to be collected includes: age, gender, race/ethnicity, stroke onset to admission, stroke types (ischemic/hemorrhagic), and stroke severity (on the National Institute of Health Stroke Severity [NIHSS] scale. Admission and discharge total Functional Independence Measure (FIM), spasticity and depression scores, ambulation velocity over 2-minutes (2-MWT) in feet/minute, and discharge disposition. The intervention is Indego® exoskeleton. The primary outcome measures were: changes in the FIM, depression and spasticity scores. The secondary outcome measure was discharge disposition. Continuous variables were analyzed using Students t-test, ordinal variables were analyzed using Mann-Whitney, and the nominal variables were analyzed using Chi-square analyses.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with acute hemorrhagic or ischemic stroke documented clinically and by neuroimaging.
2. Medically stable from a cardio-respiratory stand point so that they can participate in daily therapies.
3. Depressed patients will be included in the study
4. Patients able to stand alone
5. Patients able to provide a written informed consent, from cognitively intact patients (admission Mini Mental Scale Examination [MMSE] greater than or equal to 21).

Exclusion Criteria:

1. Aphasic patients unable to communicate
2. Confused patients
3. Patients medically unstable
4. Patients unable to stand alone
5. Refusal to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
The Functional Independence Measure (FIM™) | Baseline (Day 1) and at 4-weeks to measure change
  It measure the degree of disability as well as the progress patients make throughout their medical rehabilitation programs. FIM Scale score varies from minimum of 18 to maximum of 126. Higher score better the outcome.
The two minute walk test (2-MWT) | Baseline (Day 1) and at 4-weeks to measure change
  It assess the walking distance over two minutes while moving at a comfortable speed. using any ambulation aids (such as cane, walkers, and rollators) used in everyday life. Normal walking speed is 360 ft.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline (Day 1) and at 4-weeks to measure change
  Clinical measure of degree of spasticity. Score varies from 0=normal tome to 4=part rigid in flexion and extension. Lower the score the better the outcome.
Discharge disposition | 4-weeks
  Looks at effectiveness of rehabilitation as to how many patients are discharged home. Higher percentage 65% and above the better outcome.
The Beck Depression Inventory (BDI) | Baseline (Day 1) and at 4-weeks to measure change
  It is a 21 item self-report rating inventory measuring characteristic attitudes and symptoms of depression. It ranges in value from 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-offs are as follows: 0-9 indicates person is not depressed, 10-18 indicates mild-moderate depression, 19-29 indicates moderate-severe depression and 30-63 indicates severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Meheroz H Rabadi, MD, MRCPI, Principal Investigator — Affiliate; Oklahoma VA Health Care System
Locations (1):
- Oklahoma City VA Health Care System, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No